CLINICAL TRIAL: NCT06655610
Title: External Trigeminal Nerve Stimulation Versus Sham Stimulation for Attention Deficit Hyperactivity Disorder in Children and Adolescents Aged 7-17 Years: Study Protocol for a Pilot and Feasibility Randomized Clinical Trial
Brief Title: External Trigeminal Nerve Stimulation for Attention Deficit Hyperactivity Disorder - Feasibility Trial
Acronym: eTNS4ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Responsible Party: Principal Investigator, Ole Jakob Storebø, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2401733
Record Dates: First submitted 2024-09-04; First posted 2024-10-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: ADHD - Attention Deficit Disorder with Hyperactivity
Keywords: ADHD; Neuromodulation; External trigeminal nerve stimulation; feasibility trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active eTNS (Experimental)
  Interventions: Device: External Trigeminal Nerve Stimulation
- Sham eTNS (Sham Comparator)
  Interventions: Device: Sham device

INTERVENTIONS:
Device: External Trigeminal Nerve Stimulation — Active eTNS will be provided by applying single, bipolar pulses of 0.5 milliseconds duration at a frequency of 125 hertz, with an active period of 30 seconds on/off. Stimulation current will range from 0.2 mili ampere (mA) to 10 mA. The level of current, which is noticeable, yet within the level of comfort, will be identified for each patient by titration at baseline. Depending on the perception of stimulation, the level of current may be altered during the four weeks of treatment, by either the guardian or adolescent in control of the settings.
  Arms: Active eTNS
Device: Sham device — The stimulator and patches will be identical in appearance to the active treatment. The guardian/the adolescent will be informed to administer the device in the same fashion as with active treatment. The sham device will however be programmed to only apply stimulation for 30 seconds every hour during sleep, optimally at a frequency of maximum 2 Hz. As with the active eTNS, the sham stimulation current will range from 0.2 to 10 mA. Such settings have previously been considered to induce the sensation of a current applied to the forehead as seen with active treatment, yet without it being therapeutically effective. Stimulation will be directed through an internal resister, which ensures draining of batteries and need for recharging after each session. The manufacture of the eTNS device (Neurosigma) will oversee the programming the sham device.
  Arms: Sham eTNS

SUMMARY:
The investigators will assess the use of the Monarch eTNS device as a non-pharmacological treatment for patients aged 7 to 17 years with ADHD.

The investigators will compare the eTNS device to a sham device. Participants will use the device for four weeks during night time. During the trial, participants will receive different questionaires to assess symptoms and will also keep a logbook to record their experience with the device.

At the end of trial, the investigators will assess what the families thought of the device, and whether it is indeed feasible to further explore the effect of the device in a larger clinical trial.

DETAILED DESCRIPTION:
External trigeminal nerve stimulation (eTNS) is a non-invasive technique involving external cutaneous stimulation of the trigeminal nerve. In 2019, the Monarch eTNS device was approved as a treatment for children with attention-deficit/hyperactivity disorder (ADHD). The Monarch eTNS device is designed to be applied at home, which offers a certain level of convenience but also necessitates a high degree of compliance and acceptability from the families.

The objective of the present trial is to assess the feasibility of and pilot a larger randomized clinical trial investigating the Monarch eTNS device versus sham for patients aged 7 to 17 years with ADHD.

The investigators will conduct a parallel-group, sham-controlled, feasibility randomised clinical trial. The investigators will include 60 children and adolescents (age 7 to 17 years) diagnosed with ADHD from three clinical sites in Denmark. Patients will be randomised to 4 weeks of active versus sham eTNS. Feasibility outcomes include completion of the trial; the number of eligible participants; treatment compliance and completion. Adverse events will be monitored throughout the trial. Exploratory clinical outcomes include ADHD core symptoms (primary) and several secondary outcomes. Autonomic functions will be evaluated by means of heart rate variability, using a heart rate sensor.

This trial will evaluate the feasibility of conducting a larger randomised clinical trial investigating the use of eTNS as a home-based, non-pharmacological intervention for children and adolescents diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 17 years of age at the time of study enrollment.
* A clinical diagnosis of ADHD according to criteria for ICD-10: F90.0, F91.0, F90.8, F90.9, F98.8C. The ADHD diagnosis must be verified by the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) using The Schedule for Affective Disorders and Schizophrenia for School-aged Children (K-SADS).
* A score above 24 on the ADHD rating scale (ADHD-RS) at baseline.
* Signed informed consent from parents/legal caretakers and from the patients aged ≥ 15.

We will include treatment-naïve patients, patients who previously have received stimulant medication, and patients in stable, ongoing stimulant medication (methylphenidate or dexamphetamines/lisdexamphetamine) during the time of the trial.

Exclusion Criteria:

* Patients receiving atomoxetine and guanfacine at the time of study enrollment will be excluded all together
* Epilepsy
* Electronic or metallic implants.
* Serious mental and/or somatic diseases other than ADHD, such as:

  * Pervasive developmental disorder not including Asperger's syndrome (ICD-10 F84.0-84.4 + F84.8-84.9)
  * Schizophrenia/paranoid psychosis (ICD-10 F20-25 + F28-29)
  * Mania or bipolar disorder (ICD-10 F30 and F31)
  * Depressive psychotic disorders (ICD-10 F32.3 + F33.3)
  * Substance dependence syndrome (ICD-10 F1x.2)
  * Cardio-vascular disorders
  * Cancer
* An Intelligence quotient (IQ) below 70 measured by the Wechsler Intelligence Scale for Children
* A substantial degree of restless sleep as reported by parents or caregivers and evaluated by the physician.
* Other disabilities that may make use of Monarch problematic.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants assessed for eligibility who consent to inclusion and randomization | Four weeks
  The investigators will compare the number of eligible participants to the number of randomized participants. We will accept a difference above 50 % (95 % CI 40.2 % to 59.6 %). A larger difference can impose difficulties with recruitment in a future randomized trial.
Compliance with the intervention | Four weeks
  The investigators will calculate the number of participants fulfilling treatment. Compliance with treatment will be defined as completing the treatment in 70 % (95 % CI 57 % to 80 %) of the nights during the four weeks. Abruption of treatment can only be accepted if it happens within less than four nights in a row.
Acceptability of the intervention | Four weeks
  The acceptability of the intervention will be assessed using a semi-structured qualitative interview guide with predefined questions:
  * How did you feel about administering and controlling the device?
  * How did your child feel about receiving this type of treatment?
  * How was it for your child to receive home-treatment with the device in addition to other strategies provided by the clinic?
  * Did the intervention have any influence on the relationship between your child and the parents/siblings/school/friends?
Completion of follow up | Four weeks
  Completion of follow-up will be defined as completing the assessment of the primary exploratory clinical outcome at the end of the intervention. The number of participants with completed outcomes will be compared to the number of participants in total. If the number of participants completing this assessment is above 90 % (95 % CI 92 % to 97 %), this will be acceptable for a future full-size trial. If the number of participants completing the assessment is below 75 %, this will introduce serious problems with the interpretation of the results.
Use of concomitant treatment | Four weeks
  Any concomitant treatment or changes in medication will be assessed for each participant and subsequently evaluated for the two groups at the end of the trial.
Safety and adverse events | Four weeks
  Parents will be able to report directly to a dedicated investigators not involved in data analysis, with any concerns regarding potential adverse events or other safety issues during the trial. Adverse events will be measured by an adverse events rating scale at the end of treatment. Height, weight and vital signs will be assessed at baseline and again following the four weeks of treatment.

OTHER OUTCOMES:
ADHD core symptoms | Four weeks
  Exploratory outcome. Measured by the ADHD-IV rating scale (parent- and teacher rated) (31). Assessed at baseline, weekly, and at end of treatment
Absence from school | Four weeks
  Exploratory outcome. Measured as total hours of absence reported by logbook (parents) and through direct contact with the teachers.
Emotional liability | Four weeks
  Exploratory outcome. Measured by Conners 3 Global index, Emotional liability subscale (parent - and teacher rated)
General behavior | Four weeks
  Exploratory outcome. Measured by the Child Behavior Checklist (CBCL) (parent - and teacher rated)
Quality adjusted life years | Four weeks
  Exploratory outcome. Measured by the Child Health Utility instrument (CHU9D) (parent/self-rated)
Functional impairment | Four weeks
  Exploratory outcome. Measured by the Weiss Functional Impairment Rating Scale (WFIRS) (parent/self-rated)
Overall severity and improvement in symptoms | Four weeks
  Exploratory outcome. Measured by the Clinical Global Impressions Scale (CGI) (investigator-rated).
Behavioral and emotional difficulties | Four weeks
  Exploratory outcome. Measured by the Strengths and Difficulties Questionnaire (SDQ) (parent - and teacher rated)
Cognitive functioning | Four weeks
  Exploratory outcome. Measured by the Behavior Ratings of Individual Executive Functions (BRIEF) (parent - and teacher rated)
Sleep quality | Four weeks
  Exploratory outcome. Measured by The Children Sleep Habits Questionnaire (CSHQ) (parent - and teacher rated). Assessed at baseline, weekly and at end of treatment.
Autonomic functions | 4 weeks
  Evaluated by means of heart rate variability, using a heart rate sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Jakob Storebø, Professor, Principal Investigator — Center for Evidence-Based Psychiatry, Psychiatric Research Unit, Psychiatry Region Zealand, 4200 Slagelse, Denmark
Locations (1):
- Center for Evidence-Based Psychiatry, Psychiatric Research Unit, Psychiatry Region Zealand, 4200 Slagelse, Denmark, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edemann-Callesen H, Huus CL, Karstoft C, Bjarnadottir E, Bikic A, Jeppesen P, Martinsen OG, Pettersen FJ, Lindschou J, Juul S, Quistgaard M, Gluud C, Storebo OJ. External trigeminal nerve stimulation versus sham stimulation for attention deficit hyperactivity disorder in children and adolescents aged 7-17 years: study protocol for a pilot and feasibility randomized clinical trial. Eur Child Adolesc Psychiatry. 2025 Dec;34(12):3833-3842. doi: 10.1007/s00787-025-02786-7. Epub 2025 Jun 16. PMID 40518459